CLINICAL TRIAL: NCT06118372
Title: Safety and Tolerability of Recombinant Von Willebrand Factor Concentrate in Adult ECMO Patients With Major Bleeding: A Phase I Study
Brief Title: Recombinant vWF Concentrate and ECMO
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Michael Mazzeffi, MD, Professor of Anesthesiology, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSR230248
Record Dates: First submitted 2023-09-21; First posted 2023-11-07 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Bleeding Disorder
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Intervention Model Description: Open label non-randomized phase I trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment with recombinant vWF (Experimental): ECMO patients with major bleeding who are enrolled in the trial will receive treatment with recombinant von Willebrand Factor a single time. The dose will be 50 IU/kg and the drug will be given intravenously.
  Interventions: Drug: Recombinant von Willebrand Factor

INTERVENTIONS:
Drug: Recombinant von Willebrand Factor — Recombinant von Willebrand Factor is a drug that is currently FDA approved to treat patients with certain types of von Willebrand Disease. In the current trial it will be used to treat ECMO patients who have acquired von Willebrand syndrome.

SUMMARY:
Adult patients on extracoporeal membrane oxygenation (ECMO) frequently experience bleeding, which is in part caused by acquired von Willebrand syndrome (vWS). Prior in vitro studies have shown that the addition of recombinant von Willebrand Factor (vWF) to ECMO patient blood samples, normalizes platelet adhesion and thrombus formation. This study is a phase I study, where adult ECMO patients with refractory bleeding will be treated with recombinant vWF a single time. The primary objectives are to evaluate the safety, tolerability, and pharmacokinetics of recombinant vWF in adult ECMO patients.

DETAILED DESCRIPTION:
Coagulopathic bleeding is a common complication during ECMO. Multiple studies suggest that major bleeding occurs in 30-70% of adult ECMO patients, with higher bleeding rates in post-cardiotomy shock and veno-arterial (VA) ECMO patients. The pathophysiology of ECMO-induced coagulopathy is complex with multiple factors contributing, including loss of large VWF multimers, thrombocytopenia, increased tissue factor pathway inhibitor levels, and platelet surface glycoprotein (GP)1ba shedding. Adult ECMO patients almost universally develop acquired von Willebrand syndrome due to loss of large VWF multimers. In a study by Kalbhenn et al., acquired von Willebrand syndrome occurred within the first 6 hours of ECMO initiation in all patients (N=59) and returned to normal within 24 hours of ECMO decannulation. The loss of large VWF multimers that occurs in ECMO patients leads to poor platelet adhesion at an injury site and excess bleeding, which in some cases can become life-threatening.

In a prior observational study, the investigators found that when adult ECMO patients with acquired von Willebrand syndrome were treated with plasma-derived vWF concentrate, it increased plasma ristocetin cofactor activity (RCo), increased the RCo-VWF antigen ratio, and improved clinical hemostasis. This preliminary data suggests that use of VWF may help to reduce bleeding in ECMO patients and is safe.

Recombinant VWF has superior ultra-large multimer content, and thus it may be even better suited to treat acquired von Willebrand syndrome, which is represented by severe loss of large vWF multimers, similar to Type 2a von Willebrand disease. Further, recombinant VWF has a longer plasma half-life than plasma-derived VWF and may be safer because it contains no Factor VIII. Factor VIII activity is often supranormal during ECMO and overaccumulation of Factor VIII can increase thrombotic risk, particularly when there is blood stasis. In two prior in vitro studies, the investigators found that when recombinant VWF was added to ECMO patient blood samples, primary hemostasis/platelet adhesion returned towards normal. In a study that compared the addition of recombinant VWF to plasma-derived VWF, the investigators found that recombinant VWF improved primary hemostasis more, while having minimal impact on thrombin generation. These data suggest that recombinant VWF may be more effective in restoring primary hemostasis, and also may have a superior safety profile. The current study will investigate the safety and tolerability of recombinant VWF in adult ECMO patients with major bleeding.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (18 years or greater)
2. On extracorporeal membrane oxygenation
3. Major bleeding defined by CTCAE class 3 or greater
4. Off systemic anticoagulation for at least 4 hours

Exclusion Criteria:

1. Platelet count less than 40 x 109/L
2. International normalized ratio> 2.0
3. Fibrinogen less than 150 mg/dL
4. Current participation in another clinical trial (interventional)
5. Heparin induced thrombocytopenia (active)
6. Acute liver failure, as indicated by bilirubin >20 mg/dL or new onset hepatic encephalopathy
7. Patient or legally authorized representative unable to give informed consent
8. Allergy to recombinant von Willebrand Factor or any component of the product based on prior exposure
9. Of childbearing age and positive pregnancy test during the same hospital admission, a pregnancy test will be mandatory for all women of child-bearing age
10. Known congenital or acquired thrombophilia
11. History of deep venous thrombosis, pulmonary embolism, circuit thrombosis, disseminated intravascular coagulation (DIC), ischemic stroke, ST elevation myocardial infarction (STEMI), or arterial thrombosis in the last 3 months.
12. History of hypersensitivity to vWF concentrate
13. Known history of vWF antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Events | 30 days after treatment
  Events that 1) cause death, 2) are life-threatening, 3) cause permanent damage, 4) required intervention to prevent harm, or 5) are otherwise serious and jeopardize the patient's safety.
Area under the plasma concentration curve from zero to infinity (h × U/dL) | 96 hours after treatment
  Pharmacokinetic parameter
Plasma half-life (hours) | 96 hours after treatment
  Pharmacokinetic parameter
Mean residence time (hours) | 96 hours after treatment
  Pharmacokinetic parameter
Clearance (mL/kg per hour) | 96 hours after treatment
  Pharmacokinetic parameter
Volume at a steady state (dL/kg) | 96 hours after treatment
  Pharmacokinetic parameter
Maximum concentration (U/dL) | 96 hours after treatment
  Pharmacokinetic parameter
Time to maximum concentration (hours) | 96 hours after treatment
  Pharmacokinetic parameter
Incremental recovery ([U/dL]/[U VWF: RCo/kg] for VWF) | 96 hours after treatment
  Pharmacokinetic parameter

SECONDARY OUTCOMES:
Change in bleeding severity class | 24 hours after treatment
  The study's secondary endpoint will be any change in consensus definitions in Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 bleeding class 24 hours after treatment with Vonvendi.
Change in bleeding/drain output volume from existing surgical drains | 24 hours after treatment
  Change in total amount of bleeding/output from existing surgical drains will be a secondary study outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mazzeffi, MD, Principal Investigator — UVA
Locations (1):
- UVA Hospital, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mazzeffi M, Bathula A, Tabatabai A, Menaker J, Kaczorowski D, Madathil R, Galvagno S, Pasrija C, Rector R, Tanaka K, Herr D. Von Willebrand Factor Concentrate Administration for Acquired Von Willebrand Syndrome- Related Bleeding During Adult Extracorporeal Membrane Oxygenation. J Cardiothorac Vasc Anesth. 2021 Mar;35(3):882-887. doi: 10.1053/j.jvca.2020.06.083. Epub 2020 Jul 3. PMID 32758410
- [Result] Mazzeffi M, Hasan S, Abuelkasem E, Meyer M, Deatrick K, Taylor B, Kon Z, Herr D, Tanaka K. Von Willebrand Factor-GP1balpha Interactions in Venoarterial Extracorporeal Membrane Oxygenation Patients. J Cardiothorac Vasc Anesth. 2019 Aug;33(8):2125-2132. doi: 10.1053/j.jvca.2018.11.031. Epub 2018 Nov 22. PMID 30595484
- [Result] Mazzeffi M, Henderson R, Krause E, Rabin J, Madathil R, Chow J, Grazioli A, Meyer M, Wu Z, Tanaka K. In Vitro Comparison of Recombinant and Plasma-Derived von Willebrand Factor Concentrate for Treatment of Acquired von Willebrand Syndrome in Adult Extracorporeal Membrane Oxygenation Patients. Anesth Analg. 2022 Feb 1;134(2):312-321. doi: 10.1213/ANE.0000000000005831. PMID 34903705
- [Result] Mazzeffi M, Gonzalez-Almada A, Wargowsky R, Ting L, Moskowitz K, Hockstein M, Davison D, Levy JH, Tanaka KA. In Vitro Treatment of Extracorporeal Membrane Oxygenation Coagulopathy with Recombinant von Willebrand Factor or Lyophilized Platelets. J Cardiothorac Vasc Anesth. 2023 Apr;37(4):522-527. doi: 10.1053/j.jvca.2022.12.028. Epub 2022 Dec 30. PMID 36690556